CLINICAL TRIAL: NCT03209999
Title: Maternal Employment in Low and Middle-income Countries is Associated With Improved Infant and Young Child Feeding in Children
Brief Title: Maternal Employment in Low and Middle-income Countries and Infant Feeding
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Scott Ickes, Assistant Professor, University of Washington
Other Study IDs: UWashington
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Feeding Behavior; Maternal Health
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fomally Employed: Mother engaged in formal employment. No intervention was assigned as this is a cross sectional study.
- Informally Employed: Mother engaged in informal employment. No intervention was assigned as this is a cross sectional study.
- Non-employed: Mother neither formally or informally employed. No intervention was assigned as this is a cross sectional study.

SUMMARY:
Using cross-sectional samples from over 40 Demographic and Health Surveys, the investigators studied the association between maternal employment and 3 indicators of Infant and Young Child Feeding (IYCF): exclusive breastfeeding (EBF) among children less than 6 months old (N=39,791) and minimum diet diversity (MDD) and minimum meal frequency (MMF) (N=137,208) among children 6 to 23 months old. Mothers were categorized as formally employed, informally employed, or non-employed. The investigators first used adjusted logistic regression models to assess the associations within each country. The investigators then used meta-analysis to pool associations across all countries and by region.

DETAILED DESCRIPTION:
Data Source and Population

The investigators analyzed cross-sectional data from the Demographic and Health Surveys (DHS). DHS surveys employ standardized questionnaires and nationally representative, multi-stage cluster sampling to allow for cross-country comparisons (34).

Our study included DHS datasets that were administered between 2010 and April 2017 and that contained data on women's employment status and indicators of IYCF. Analyses included women who had at least one child between ages 0-24 months. If mothers had more than one child, the investigators included the youngest child in the household. Children residing outside the household were excluded.

In models that evaluated MDD and MMF as the dependent variables, the final analytic sample included 137,208 children aged 6 to 23 months from 50 countries. Small cell sizes were prohibitive to exploring the employment-EBF associations in 10 countries that met the aforementioned inclusion criteria; therefore, when modeling EBF as the dependent variable, the final analytic sample included 39,791 children aged 0 to 5 months in 40 countries.

Primary Dependent Variables

EBF, MDD, and MMF served as the primary dependent variables of interest as prior literature suggests changes in women's income and time, stemming from women's employment, may affect these indicators of IYCF. These indicators were created using data from the 24-hour recall of foods/food groups available in DHS. EBF, a binary variable, was defined as the proportion of infants 0 to 5 months of age who were fed exclusively with breast milk. MDD, a binary variable, was defined as proportion of children 6 to 23 months of age who received foods from 4 or more of the following 7 food groups: grains, roots and tubers; legumes and nuts; dairy products (milk, yogurt, cheese); flesh foods (meat, fish, poultry and liver/organ meats); eggs; vitamin-A rich fruits and vegetables; and other fruits and vegetables. MMF, a binary variable, was defined as the proportion of breastfed and non-breastfed children 6 to 23 months of age who receive solid, semi-solid, or soft foods the minimum number of times or more. For breastfed children, the minimum number of times varies with age (2 times if 6 to 8 months and 3 times if 9 to 23 months). Non-breastfed children ages 6 to 23 months must be fed 4 or more times per day to meet the MMF indicator.

Primary Independent Variable

The investigators modeled maternal employment as a 3-category variable: formally employed, informally employed, and non-employed based on prior research which suggests: 1) a large proportion of women in LMIC are engaged in less formalized employment and 2) wages earned are more than 60% lower in the informal sector. Women are described as non-employed because this term includes persons who choose to not seek employment whereas unemployed describes persons without jobs who are actively seeking employment.

Employment type was defined based on 4 indicators: 1) employment status in the last 12 months (employed, non-employed); 2) aggregate occupation category (skilled, unskilled); 3) type of earnings (cash only, cash and in-kind, in-kind only, unpaid); and 4) seasonality of employment (all year, seasonal/occasional employment). Formal employment included the following 3 combinations: 1) employed, skilled occupation, cash only earnings, employed all year; 2) employed, skilled occupation, cash only earnings, seasonal/occasional employment; and 3) employed, unskilled occupation, cash only earnings, employed all year. Other employed women were categorized as informally employed.

Confounders and Effect Measure Modifiers

The investigators identified confounding factors a priori using a directed acyclic graph, which is a causal diagram used to characterize the relationship among variables that influence the primary independent and the dependent variables based on both theorized and documented relationships. In all models, confounders included maternal education (< primary school complete, [Symbol] primary school complete), maternal age (years), marital status (married or living together versus single, widowed, divorced), parity, morbidity (presence of diarrhea or fever in the last two weeks), child age (months), and urban/rural status. The investigators aimed to specify covariates in a way that allowed for the same specification in each country and for each outcome. For variables that were in their continuous form in the DHS (maternal age, child age, parity), the investigators assessed their linearity with the outcomes by specifying disjoint indicator variables. Because variables were approximately linearly associated with the outcomes in most countries, they were retained in their continuous form to minimize the number of observations dropped from the model due to small cell sizes. Marital status and maternal education were dichotomized because there were very few people in some categories (e.g. divorced).

The investigators hypothesized that the employment-diet association would vary by countries' stage in the nutrition transition. Therefore, the investigators explored differences in the country-level associations by log-gross domestic product (GDP) per capita, adjusted for purchasing power parity, a theorized driver of the nutrition transition (41). Data were obtained from the World Development Indicators database, corresponding to the survey year (42). GDP-per capita was log-transformed to reflect the expected influence of a percent increase (e.g. 5%), rather than an absolute dollar increase (e.g. $5).

Statistical Analysis

Within-country analyses. It is expected that trends in employment (i.e. the percent of women in formal versus informal employment) as well as diet to differ depending on countries' stage of the nutrition transition. Therefore, the investigators aimed to keep samples comparable by selecting countries with a recent DHS (2010-2017) and we allowed for different relationships in each country by starting with disaggregate, country-specific estimates. The investigators first employed separate multivariable logistic regression models for each country to test the association between maternal employment and IYCF indicators (EBF, MDD, MMF). In these country-specific models, the investigators utilized sampling weights to account for differential probability of selection and response and Taylor series linearized standard errors accounted for DHS' clustered design.

Between-country and region analyses. After obtaining disaggregated estimates for each country, coefficients for the employment-EBF, employment-MDD, and employment-MMF associations were entered into a random effects meta-analysis to obtain odds ratios pooled across all countries and by world region (East Asia and Pacific, Europe and Central Asia, Latin American and Caribbean, Middle East and North Africa, South Asia, and sub-Saharan Africa). Random effects meta-analysis, used to generate pooled odds ratios (POR), is the statistical combination of the estimates from separate countries and assumes that the associations between employment and IYCF may differ by country and/or region.

Country-specific beta coefficients were also entered into a random-effects meta-regression to assess whether the associations between employment and IYCF varied by country-level log-GDP.

Sensitivity Analyses. Sensitivity analyses included modeling several alternative outcomes including: 1) continued breastfeeding at 1 year, 2) diet diversity score, and 3) minimum acceptable diet. Continued breastfeeding at 1 year, a binary variable, was defined as the proportion of children 12 to 15 months of age who are fed breast milk (37). Diet diversity score, a continuous variable estimated among children aged 6 to 23 months, was based on the aforementioned 7 foods groups used to calculate MDD (37). For each of the 7 food groups, children received 1 point if any food in the group was consumed (i.e. minimum DDS =0, maximum DDS =7). Minimum acceptable diet was modeled as a binary variable and was defined as the proportion of children 6 to 23 months of age who received a minimum acceptable diet as determined by minimum food frequency, diet diversity, and breastfeeding status (37). Because in some cases the within-country sample size for the associations between employment and EBF were somewhat smaller, we also employed a single logistic regression model with all 40 countries to test the association between employment and EBF. In this specification, each country was included as a fixed-effect, and therefore controlled for baseline country-level differences; but this model assumes the association between employment and EBF is homogeneous across countries. Alpha was set to 0.05. Analyses were performed using Stata 14.1 (StataCorp LP, College Station, Texas). No institutional review board review was obtained given that all analyses used secondary data.

ELIGIBILITY:
Inclusion Criteria:

* Last born child, ages 1 to < 24 months
* Child living with mother

Exclusion Criteria:

* Complete data available for maternal employment, children's dietary diversity, minimum meal frequency data
* Complete covariates available for maternal education, maternal age, marital status, parity, morbidity in the past 2 weeks, child age, and urban/rural status

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Maternal-child dyads within one of 50 low and middle-income countries with a Demographic and Health Survey since 2010
Sampling Method: Non-Probability Sample
Enrollment: 39791 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Exclusive Breastfeeding | 0 to 6 months
  Prevalence odds of exclusive breastfeeding among children under 6 months

SECONDARY OUTCOMES:
Minimum Dietary Diversity | 6 to 23 months
  Prevalence odds of minimum dietary diversity among children 6 to 23 months
Minimum Meal Frequency | 6 to 23 months
  Prevalence odds of minimum meal frequency among children 6 to 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Ickes, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oddo VM, Ickes SB. Maternal employment in low- and middle-income countries is associated with improved infant and young child feeding. Am J Clin Nutr. 2018 Mar 1;107(3):335-344. doi: 10.1093/ajcn/nqy001. PMID 29566201